CLINICAL TRIAL: NCT03476785
Title: Prevention of Cardiovascular Stiffening With Aging and Hypertensive Heart Disease
Acronym: LVH
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Texas Southwestern Medical Center (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: STU 062014-068
Record Dates: First submitted 2018-03-01; First posted 2018-03-26 (Actual); Last update posted 2019-10-14 (Actual); Status verified 2019-10

CONDITIONS: Lv Hypertrophy; Heart Failure, Diastolic; Stiffness, Vascular
Keywords: LVH; Ventricular Stiffness; Fitness; HFpEF
MeSH Terms: conditions — Hypertrophy, Left Ventricular; Heart Failure, Diastolic | interventions — High-Intensity Interval Training; Yoga

STUDY DESIGN:
Intervention Model Description: Parallel Assignment
Who Masked: Outcomes Assessor
Masking Description: Outcomes assessor will be blinded to subject randomization.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- High Intensity Exercise (Experimental): Subjects randomized to receive high intensity aerobic exercise will undergo exercise training for 1 year. A training program will be developed individually for each subject with the goal of increasing duration and intensity consistent with exercise training principles. Workouts will vary with respect to mode (walk, cycle) and duration (30 - 60 minutes). Each subject will be assigned an exercise physiologist and a heart rate monitor so that each session can be tracked and recorded.
  Interventions: Behavioral: High intensity exercise
- Yoga (Placebo Comparator): Subjects randomized to yoga will receive instructions on strength and flexibility exercises.
  Interventions: Behavioral: Yoga

INTERVENTIONS:
Behavioral: High intensity exercise — Subjects will perform high intensity aerobic exercise in addition to moderate intensity sessions 4-5 times per week.
  Arms: High Intensity Exercise
Behavioral: Yoga — Subjects will perform strength and flexibility exercises.
  Arms: Yoga

SUMMARY:
The purpose of this study is to determine whether vigorous exercise training 4-5 days/week for one year in sedentary middle aged (ages 40-64) individuals at high risk for future development of heart failure will improve cardiac and vascular compliance to a degree equivalent to life-long exercisers and the sedentary young. To date, no effective therapy for heart failure with preserved ejection fraction (HFpEF) has been found; therefore prevention is critical and discovering novel treatment strategies is essential. Exercise training if implemented in high risk patients may improve diastolic function and cardiac-vascular interactions, preventing further progression to overt heart failure.

DETAILED DESCRIPTION:
The global objective of this project is to test novel strategies to prevent diastolic dysfunction associated with HFpEF; these include: a) identifying high risk individuals by using population derived imaging and blood biomarkers; and b) implementing novel exercise training strategies in these middle age individuals, when cardiac plasticity still exists, to forestall the development of diastolic abnormalities that progress to HFpEF.

Prior research has demonstrated that: a) healthy but sedentary aging leads to atrophy and stiffening of the heart with reduced myocardial and chamber compliance; b) in contrast, highly competitive senior athletes had cardiac compliance that was indistinguishable from healthy young individuals suggesting that lifelong exercise training prevented this stiffening; c) even prolonged and intense exercise training started after age 65 failed to reverse age-related cardiac and vascular stiffening; d) cardiac stiffening begins in middle age (40-64) and can be substantially prevented by training 4-5 days/wk. The primary objective of this project is therefore to identify high risk sedentary individuals age 40-64, and initiate an exercise program carefully designed to maximize effects on cardiovascular compliance and function. Findings from this aim would have enormous public health significance and establish a novel, practical exercise training strategy designed to reverse cardiovascular stiffening.

Hypothesis:

Exercise training, when implemented 4-5 times/week over a prolonged period of time in sedentary high risk middle aged men and women, age 40-64 will improve cardiac and vascular compliance to a degree equivalent to life-long exercisers (and sedentary young);

Specific Aim:

To test the hypothesis, two groups of previously sedentary subjects, ages 40-64 at particularly high risk for HF will be studied for one year, with the following interventions: 1) subjects undergoing prolonged endurance/interval/strength exercise training; and 2) strength and flexibility /balance control. Subjects will be categorized as high risk and enrolled on the basis of elevated serum biomarkers and left ventricular hypertrophy (LVH) documented by cardiac MRI. Comprehensive invasive and non-invasive assessment of cardiovascular structure and systolic/diastolic function will be performed before and after 1 year of an exercise intervention involving high intensity aerobic intervals, lower intensity endurance training, and strength training, compared with strength and flexibility control.

ELIGIBILITY:
Inclusion Criteria:

* Presence of left ventricular hypertrophy (by MRI, echocardiography or ECG)
* Normal ejection fraction (>50%)
* Elevated cardiac biomarker (high sensitivity troponin, NT-BNP)

Exclusion Criteria:

* age < 40 or >64
* body mass index>35
* history of heart failure, myocarditis, restrictive cardiomyopathy, severe chronic obstructive pulmonary disease, unstable coronary artery disease or recent (<12 month) acute coronary syndrome, cerebrovascular disease as evidenced by prior transient ischemic attack or stroke and active/recent tobacco use (quit < 5 years).
* chronic orthopedic injury that precludes exercise testing

Ages: 40 Years to 64 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 56 (Actual)
Dates: Start 2015-06-01 (Actual); Primary Completion 2019-07-02 (Actual); Study Completion 2019-07-02 (Actual)

PRIMARY OUTCOMES:
Left ventricular stiffness | 1 year
  Change in ventricular stiffness after 1 year of exercise training measured as the stiffness constant of the diastolic limb of the left ventricular pressure-volume curve

SECONDARY OUTCOMES:
Aerobic fitness | 1 year
  Change in peak aerobic capacity (VO2) after 1 year of exercise training
Vascular stiffness | 1 year
  Change in pulse wave velocity after 1 year of exercise training

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin D Levine, MD, Principal Investigator — University of Texas Southwestern Medical Center
Locations (1):
- The Institute for Exercise and Environmental Medicine, Dallas, Texas, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Hieda M, Sarma S, Hearon CM Jr, MacNamara JP, Dias KA, Samels M, Palmer D, Livingston S, Morris M, Levine BD. One-Year Committed Exercise Training Reverses Abnormal Left Ventricular Myocardial Stiffness in Patients With Stage B Heart Failure With Preserved Ejection Fraction. Circulation. 2021 Sep 21;144(12):934-946. doi: 10.1161/CIRCULATIONAHA.121.054117. Epub 2021 Sep 20. PMID 34543068
- [Derived] Hieda M, Sarma S, Hearon CM Jr, Dias KA, Martinez J, Samels M, Everding B, Palmer D, Livingston S, Morris M, Howden E, Levine BD. Increased Myocardial Stiffness in Patients With High-Risk Left Ventricular Hypertrophy: The Hallmark of Stage-B Heart Failure With Preserved Ejection Fraction. Circulation. 2020 Jan 14;141(2):115-123. doi: 10.1161/CIRCULATIONAHA.119.040332. Epub 2019 Dec 23. PMID 31865771